CLINICAL TRIAL: NCT01384539
Title: Vitamin D and Arterial Function in Patients With Chronic Kidney Disease
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 11-0521; 5K23DK087859 (NIH)
Record Dates: First submitted 2011-06-27; First posted 2011-06-29 (Estimated); Results first posted 2017-08-17 (Actual); Last update posted 2018-09-28 (Actual); Status verified 2018-08

CONDITIONS: Arterial Dysfunction; Chronic Kidney Disease
Keywords: chronic kidney disease; vitamin D deficiency
MeSH Terms: conditions — Renal Insufficiency, Chronic; Vitamin D Deficiency | interventions — Cholecalciferol; Calcitriol

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cholecalciferol (Experimental): Cholecalciferol 4000 IU capsule by mouth daily x 1 month then 2000 IU capsule by mouth daily x 5 months
  Interventions: Drug: Cholecalciferol
- Calcitriol (Experimental): Calcitriol 0.25 mcg capsule by mouth daily x 1 month then 0.5 mcg capsule by mouth daily x 5 months
  Interventions: Drug: Calcitriol

INTERVENTIONS:
Drug: Cholecalciferol
  Arms: Cholecalciferol
Drug: Calcitriol
  Arms: Calcitriol

SUMMARY:
The purpose of this study is to determine whether nutritional (cholecalciferol) or active vitamin D (calcitriol) supplementation improves vascular endothelial function in patients with stage IIIB and IV chronic kidney disease with vitamin D insufficiency or deficiency. The investigators hypothesize that the use of calcitriol supplementation will result in improved vascular endothelial function as compared to cholecalciferol supplementation.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Chronic kidney disease stage IIIB or IV by 4 parameter Modified Diet in Renal Diseases Formula (Estimated Glomerular Filtration Rate [GFR] 44-15 ml/min/1.73m2)
* Vitamin D (D2 + D3) deficient, defined as serum 25(OH)D level < 30 ng/mL
* Corrected serum calcium < 10.2 mg/dL
* Serum phosphate < 4.6 mg/dL
* Serum albumin > 3.0 g/dL
* Body mass index < 40 kg/m2
* Ability to give informed consent

Exclusion Criteria:

* Significant co-morbid conditions that lead the investigator to conclude that life expectancy is less than 1 year
* Expected to undergo living related kidney transplant in next 6 months
* Pregnant, breastfeeding, or unwilling to use adequate birth control
* History of severe liver disease
* Nephrotic range proteinuria (> 3.5 gm/day)
* Use of active vitamin D analogs within 30 days of randomization

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 128 (Actual)
Dates: Start 2011-07 (Actual); Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jessica Kendrick, MD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado Denver Clinical Translational Research Center, Aurora, Colorado, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Cholecalciferol: Cholecalciferol 4000 IU capsule by mouth daily x 1 month then 2000 IU capsule by mouth daily x 5 months
  Cholecalciferol
- Calcitriol: Calcitriol 0.25 mcg capsule by mouth daily x 1 month then 0.5 mcg capsule by mouth daily x 5 months
  Calcitriol
Period: Overall Study
Arm/Group | Cholecalciferol | Calcitriol
Started | 64 | 64
Completed | 58 | 57
Not Completed | 6 | 7

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Cholecalciferol | Calcitriol | Total
Number analyzed (Participants) | 64 | 64 | 128
Age, Continuous [Mean (Standard Deviation); unit: years] | 58 (13) | 59 (12) | 58 (12)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19 | 23 | 42
  Male | 45 | 41 | 86
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Non-Hispanic White | 23 | 23 | 46
  Non-Hispanic Black | 18 | 14 | 32
  Hispanic | 16 | 23 | 39

OUTCOME MEASURES:

1. Primary Outcome: Compare the Difference Between the Calcitriol and Cholecalciferol Groups in Conduit Artery Endothelium-dependent Dilation (EDD) in Response to Treatment.
Description: EDD will be measured by brachial artery flow-mediated dilation (FMD). The mean change in percent FMD from baseline will be documented.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: percent change in FMD
Arm/Group | Cholecalciferol | Calcitriol
Number analyzed (Participants) | 58 | 57
percent change in FMD | -0.5 (4.2) | 0.3 (3.5)

2. Secondary Outcome: Compare the Efficacy of Calcitriol and Cholecalciferol Supplementation on Plasma Concentrations of C-reactive Protein
Description: Secondary aims are focused to explore whether vitamin D improves vascular endothelial function through decreases in inflammation
Time Frame: 6 months
Measure: Median (Inter-Quartile Range); unit: mg/dL
Arm/Group | Cholecalciferol | Calcitriol
Number analyzed (Participants) | 58 | 57
mg/dL
  Baseline | 3.0 [1.2 to 7.9] | 3.4 [1.5 to 6.7]
  End of Study | 3.1 [1.7 to 8.3] | 3.9 [0.3 to 2.1]

3. Secondary Outcome: Compare the Effect of Calcitriol and Cholecalciferol Supplementation on Vascular Endothelial Cell Expression of Nf-kB
Description: The effect of calcitriol and cholecalciferol supplementation will be evaluated calculating the mean change in total vascular endothelial cell NFkB expression. NFkB expression is given as arbitrary units and represent ratios of endothelial cell protein expression to human umbilical vein endothelial cell (HUVEC) expression in order to account for any variation in the staining procedure.
Time Frame: 6 months
Measure: Mean (Standard Deviation); unit: ratio of NFkB to HUVEC expression
Arm/Group | Cholecalciferol | Calcitriol
Number analyzed (Participants) | 58 | 57
ratio of NFkB to HUVEC expression | 0.03 (0.1) | -0.01 (0.1)

ADVERSE EVENTS:
Arm/Group | Cholecalciferol | Calcitriol
All-Cause Mortality (participants affected / at risk) | 2/64 | 0/64
Serious Adverse Events (participants affected / at risk) | 9/64 | 5/64
Other Adverse Events (participants affected / at risk) | 1/64 | 4/64
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol (N=64) | Calcitriol (N=64)
Hospitalization (Cardiac disorders) | 9 (9) | 5 (5) — Hospitalization for congestive heart failure, myocardial infarction, stroke, and/or angina
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Cholecalciferol (N=64) | Calcitriol (N=64)
Hypercalcemia (Renal and urinary disorders) | 1 (1) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No